CLINICAL TRIAL: NCT05240404
Title: A Randomized Phase II Study of Adjuvant Immunotherapy With Toripalimab Following Curative-intent Ablation for Recurrent Hepatocarcinoma
Brief Title: Adjuvant Immunotherapy With Toripalimab Following Curative-intent Ablation for Recurrent Hepatocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRTOE
Record Dates: First submitted 2022-02-07; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Immunotherapy; Toripalimab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab; Immunotherapy; Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): Patients with recurrent hepatocellular carcinoma would be treated with curative-intent ablation alone.
  Interventions: Procedure: Thermal ablation
- Arm B (Experimental): Patients with recurrent hepatocellular carcinoma would be treated with curative-intent ablation and adjuvant immunotherapy with toripalimab.
  Interventions: Drug: Toripalimab; Procedure: Thermal ablation

INTERVENTIONS:
Drug: Toripalimab — toripalimab treatment (240mg intravenously every 3 weeks) started on day 3 after ablation for six months
  Other Names: Immunotherapy
  Arms: Arm B
Procedure: Thermal ablation — The ablation operation was performed under local or compound anesthesia and guided by ultrasonography (US) or computed tomography (CT). To ensure complete destruction of the tumor, the ablation area must exceed the tumor boundary 1.0 cm.
  Other Names: Local treatment

SUMMARY:
This phase II study is to evaluate the efficacy of the adjuvant immunotherapy after curative-intent ablation for recurrent hepatocarcinoma

ELIGIBILITY:
Inclusion Criteria:

HCC diagnosed as (i) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level greater than 200 IU/ml and a radiologically compatible feature with HCC in one or more CT/MRI/angiograms, or (ii) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level less than 200 IU/ml, and a radiologically compatible feature with HCC in two or more CT/MRI/angiograms or (iii) histological confirmation.

HCC patients who had recurrent or residual tumor after other treatments without evidence of extrahepatic metastasis the largest diameter of tumor should be less than 3cm, and the number of tumor ≤2 no previous treatment to target tumors by other forms of RT.

liver function of Child-Pugh class A or B7 (Child-Pugh score of ≤7). performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score.

WBC count ≥ 2,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 50,000/mm3; and adequate hepatic function (total bilirubin ≤ 3.0 mg/dL; AST and ALT < 5.0× upper limit of normal; no ascites).

no serious comorbidities other than liver cirrhosis. written informed consent.

Exclusion Criteria:

HCC diagnosed as (i) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level greater than 200 IU/ml and a radiologically compatible feature with HCC in one or more CT/MRI/angiograms, or (ii) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level less than 200 IU/ml, and a radiologically compatible feature with HCC in two or more CT/MRI/angiograms or (iii) histological confirmation.

HCC patients who had recurrent or residual tumor after other treatments without evidence of extrahepatic metastasis the largest diameter of tumor should be less than 3cm, and the number of tumor ≤2 no previous treatment to target tumors by other forms of RT.

Liver function of Child-Pugh class A or B7 (Child-Pugh score of ≤7). Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score.

WBC count ≥ 2,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 50,000/mm3; and adequate hepatic function (total bilirubin ≤ 3.0 mg/dL; AST and ALT < 5.0× upper limit.

Written informed consent.

Exlusion criteria:

Evidence of extrahepatic metastasis. Liver function of Child-Pugh class B8-9 and C (Child-Pugh score of >7). Previous history of other forms of RT adjacent to target tumors. Poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score.

Pregnant or breast feeding status. Previous history uncontrolled other malignancies within 2 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | up to 3 years until study closed
  Disease-free survival was defined as the interval from the date of randomization to date of detection new recurrent disease

SECONDARY OUTCOMES:
Overall survival | up to 3 years until study closed
  Overall survival (OS) was defined as the interval from the date of randomization to death or study closed
Number of participants with adverse events | Up to approximately 3 years
  Evaluation will be done using NCI-CTCAE (version 4.03).
Predictive Biomarkers | Up to approximately 3 years
  Tissue and blood biomarkers in including PD-L1 expression, tumor mutation burden defined as the number of non-inherited mutations per million bases of investigated genomic sequence

CONTACTS AND LOCATIONS:
Overall Officials: Liangrong Shi, M.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China